CLINICAL TRIAL: NCT06904599
Title: Evaluation of Human Chorionic Gonadotropin for the Treatment of Acute Graft-versus-host Disease in Patients With Allogeneic Hematopoietic Cell Transplantation
Brief Title: Efficacy of Human Chorionic Gonadotropin in Acute GVHD Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Collaborators: Marisa Romero Martínez (Unknown); Dr. José Carlos Jaime Perez (Unknown); Dr. David Gómez Almaguer (Unknown); Dra. Consuelo Mancias Guerra (Unknown); Dr. Andrés Gómez de León (Unknown); Dra. Olga Graciela Catú Rodríguez (Unknown); Dra. Perla Colunga Pedraza (Unknown); Dra. Michelle Morcos Sandino (Unknown)
Responsible Party: Principal Investigator, Cesar Homero Gutierrez-Aguirre, Principal Investigator, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE25-00006
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Acute Graft Versus Host Disease
Keywords: Acute GVHD; human chorionic gonadotropin
MeSH Terms: interventions — Chorionic Gonadotropin; Prednisone; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Clinical, longitudinal, prospective, phase 2, randomized, comparative, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Active Comparator): Oral prednisone 1 mg/kg/day for 14 days or IV dexamethasone 0.15 mg/kg/day for 14 days + human chorionic gonadotropin 2500 IU intramuscular on days 1, 3, and 5 of the protocol. Patients who have at least a partial response by day 7 will receive 3 weekly doses for an additional 4 weeks.
  Interventions: Drug: Human chorionic gonadotropin (hCG); Drug: Prednisone; Drug: Dexamethasone
- Control group (Active Comparator): Oral prednisone 1 mg/kg/day for 14 days or IV dexamethasone 0.15 mg/kg/day for 14 days.
  Interventions: Drug: Prednisone; Drug: Dexamethasone

INTERVENTIONS:
Drug: Human chorionic gonadotropin (hCG) — 2500 IU intramuscular on days 1, 3, and 5 of the protocol. Patients who have at least a partial response by day 7 will receive 3 weekly doses for an additional 4 weeks.
  Arms: Study group
Drug: Prednisone — Oral prednisone 1 mg/kg/day for 14 days
Drug: Dexamethasone — IV dexamethasone 0.15 mg/kg/day for 14 days

SUMMARY:
Graft-versus-host disease is a complication of allogeneic hematopoietic cell transplantation with high morbidity and mortality. The standard treatment is corticosteroids, and based on the response within 3 to 7 days, a second-line therapy is added, which is expensive and not easily accessible. The administration of human chorionic gonadotropin has shown therapeutic effectiveness in 50% of patients in reported clinical cases.

DETAILED DESCRIPTION:
The study will include 20 patients with recent-onset allogeneic hematopoietic cell transplantation and GVHD who attend the Hematology Service at the University Hospital and meet the inclusion criteria, to receive conventional treatment with steroids (prednisone 1 mg/kg/day for 14 days) or combined treatment (hCG 2500 IU, IM + prednisone 1 mg/kg/day for 14 days).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Any gender.
* Post-allogeneic transplantation status (haploidentical or identical) of hematopoietic cells.
* Presenting recently onset aGVHD, grades 2 to 4, and requiring systemic steroid use as determined by the treating physician.
* Have not received steroids (Prednisone ≥1 mg/kg/day or equivalent dose of another steroid) for more than 3 days in the last week.
* Willing to participate in the study by signing informed consent.
* If the subject is female and has the potential to procreate (a woman is considered fertile from menarche to postmenopausal stage or after undergoing a permanent contraceptive method), she agrees to use one of the following contraceptive methods from the start of the study and for 30 days after the protocol: oral hormonal contraception, intrauterine device, barrier methods (diaphragm, male or female condom, and foam, sponge, or spermicide film), or agrees to remain abstinent. Women who have been postmenopausal for more than a year, undergone hysterectomy, bilateral oophorectomy, or bilateral salpingectomy are not considered to have reproductive potential.
* If the subject is male, he agrees to use one of the following contraceptive methods from the start of the study and for 30 days after the protocol: male condom, or remain abstinent.

Exclusion Criteria:

* Arterial or venous thrombosis in the past 3 months.
* History of thromboembolic disease requiring full-dose anticoagulation.
* Diagnosis of active malignant disease.
* Uncontrolled infection.
* Chronic use of supplemental therapy with sex hormones (estrogen, progesterone, and/or testosterone).
* Women with a positive pregnancy test at the time of the initial evaluation.
* Women or men of reproductive age who are unwilling to take appropriate precautions to avoid an unwanted pregnancy from the start of the protocol until 30 days after the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of GVHD response | 1 year
  The primary outcome measure for this study is the effectiveness of human chorionic gonadotropin (hCG) when combined with steroids in the treatment of acute graft-versus-host disease (aGVHD) in patients with allogeneic hematopoietic cell transplantation (allo-HCT). This could be assessed using clinical criteria such as improvement in skin, liver, gastrointestinal symptoms, and overall patient condition, evaluated at specified time points (e.g., day 7, day 14, and at the end of the treatment regimen).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.nature.com/articles/bmt2015220
- See also: Related Info — https://www.nature.com/articles/bmt201459